CLINICAL TRIAL: NCT00286364
Title: Short-Term Androgen Priming Before COS Using Aromatase Inhibitor and hCG During Early-Follicular-Phase GnRH Antagonist Administration - a Randomized Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: version 01.2005-05-20; NCT00150501 (obsolete NCT alias)
Record Dates: First submitted 2006-02-01; First posted 2006-02-03 (Estimated); Last update posted 2007-04-23 (Estimated); Status verified 2007-04

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Down-Regulation; Aromatase Inhibitors

INTERVENTIONS:
Drug: Downregulation and androgen priming by use of GnRH antagonist, aromatase inhibitor and hCG before COH

SUMMARY:
We want to investigate if early follicular phase downregulation and androgen priming, by use of GnRH antagonist, aromatase inhibitor and hCG before COH in a short protocol, shows signs of improvement compared to standard short antagonist protocol

ELIGIBILITY:
Inclusion Criteria:

* Indication and wish for IVF/ICSI treatment
* Womens age 20-39 years (both inclusive)
* Regular menstrual cycle within normal range
* Body Mass Index: 18-30 kg/m2 (both inclusive)
* Negative pregnancy test before treatment
* A maximum of 3 earlier IVF/ICSI treatments that did not result in pregnancy

Exclusion Criteria:

* serious systemic disease
* Presence of polycystic ovarian syndrome (PCOS)
* Earlier poor response with less than 4 mature follicles
* Earlier participation in the investigation

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Lossl, medical doctor, Principal Investigator — The Fertility Clinic 4071, Copenhagen University Hospital Rigshospitalet
Locations (1):
- The Fertility Clinic 4071, Copenhagen University Hospital Rigshospitalet, Copenhagen, Copenhagen East, Denmark

REFERENCES:
- [Derived] Lossl K, Andersen CY, Loft A, Freiesleben NL, Bangsboll S, Andersen AN. Short-term androgen priming by use of aromatase inhibitor and hCG before controlled ovarian stimulation for IVF. A randomized controlled trial. Hum Reprod. 2008 Aug;23(8):1820-9. doi: 10.1093/humrep/den131. Epub 2008 May 15. PMID 18487212